CLINICAL TRIAL: NCT04067258
Title: Evaluation of Choroidal Thickness in Patients Suffering From Beta-thalassemia
Brief Title: Choroidal Thickness in Beta-thalassemia Patients
Status: Completed | Type: Observational
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Associate Professor in Ophthalmology, University Hospital of Patras
Other Study IDs: 9894 / 20 -5 -2016
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Beta-Thalassemia
Keywords: beta-thalassemia; choroidal thickness; enhanced depth imaging; optical coherence tomography
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Beta-Thalassemia group: Patients suffering from beta thalassemia major or intermedia will be included in this group
  Interventions: Diagnostic Test: EDI-OCT
- Control group: Healthy age and sex matched volunteers will be included in this group
  Interventions: Diagnostic Test: EDI-OCT

INTERVENTIONS:
Diagnostic Test: EDI-OCT — EDI-OCT (enhanced depth imaging spectral domain optical coherence tomography) wiil be performed in all study participants.
  Three sets of measurements in the macular (horizontal and vertical) and peripapillary area will be averaged.

SUMMARY:
The purpose of this study is to examine choroidal thickness in beta-thalassemia patients and compare it to the one of healthy controls.

An equal number of transfusion dependent beta-thalassemic patients and age and sex matched healthy volunteers will undergo spectral-domain optical coherence tomography utilizing the enhanced depth imaging application to visualize and measure the choroid.

DETAILED DESCRIPTION:
Beta thalassemia is an inherited hemoglobinopathy, associated with defective production of beta-chain globin resulting in problematic HbA production. It is classified according to the severity as minor, intermedia and major. Patients suffering from beta-thalassemia intermedia and beta-thalassemia major require regular blood transfusions. Transfusion related hemosiderosis in these patients necessitates the use of chelating agents to prevent iron overload in vital organs such as the liver and heart.

A number of ocular abnormalities can present in beta-thalassemia patients. Those are categorized as pseudoxanthoma elasticum (PXE)-like changes that include angioid streaks, peau d'orange like fundus and optic nerve head drusen and non-PXE-like changes such as increased venous tortuosity.

Furthermore, it is well established that prolonged treatment with some of the chelating agents such as deferoxamine are associated with ocular toxicity, namely nyctalopia, colour perception anomalies, visual field disturbances, cataract formation, optic neuropathy and pigmentary retinopathy.

The pathophysiology of those ocular manifestations has not been fully clarified. The role of the choroid has not been determined since this particular tissue was previously unaccessible to imaging. Enhanced depth imaging optical coherence tomography is able to image the choroid providing reasonable clarity compared to spectral domain optical coherence tomography.

The aim of this study is to evaluate possible alterations of choroidal thickness in beta thalassemia as compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Beta thalassemia patients undergoing blood transfusions

Exclusion Criteria:

* History of glaucoma, keratoconus, retinal disease, ocular trauma, ocular surgery, uveitis, amblyopia, strabismus, ocular vascular abnormalities
* Spherical refractive error greater than 4 diopters or cylindrical refractive error greater than 2 diopters
* History of other systemic disease such as uncontrolled hypertension, diabetes mellitus, or connective tissue disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with beta-thalassemia major or intermedia undergoing blood transfusions will be examined utilizing EDI-OCT.
  A group of equal healthy volunteers will also be included to serve as controls.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Subfoveal choroidal thickness | 8-10 am
  Manual measurements of the choroid starting from the end of the retinal pigment epithelium throughout the outline of the sclera, will be conducted subfoveally

SECONDARY OUTCOMES:
Choroidal thickness nasally to the fovea | 8-10 am
  Manual measurements of the choroid starting from the end of the retinal pigment epithelium throughout the outline of the sclera, will be conducted at anatomic locations nasally to the subfoveal point
Choroidal thickness inferiorly to the fovea | 8-10 am
  Manual measurements of the choroid starting from the end of the retinal pigment epithelium throughout the outline of the sclera, will be conducted at anatomic locations inferiorly to the subfoveal point
Choroidal thickness temporally to the fovea | 8-10 am
  Manual measurements of the choroid starting from the end of the retinal pigment epithelium throughout the outline of the sclera, will be conducted at anatomic locations temporally to the subfoveal point
Choroidal thickness superiorly to the fovea | 8-10 am
  Manual measurements of the choroid starting from the end of the retinal pigment epithelium throughout the outline of the sclera, will be conducted at anatomic locations superiorly to the subfoveal point
Peripapillary choroidal thickness (inferior, superior, nasal and temporal fields) | 8-10 am
  Manual measurements of the choroid starting from the end of the retinal pigment epithelium throughout the outline of the sclera, will be conducted at the inferior, superior, nasal and temporal quadrants in the peripapillary area.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, General University Hospital of Patras, Pátrai, Achaea, Greece